CLINICAL TRIAL: NCT05807412
Title: A Prospective, Single-center, Blinded, Randomized, Split-face Study Evaluating the Spread of PrabotulinumtoxinA-xvfs Versus OnabotulinumtoxinA in the Treatment of Forehead Rhytides
Brief Title: Spread of PrabotulinumtoxinA-xvfs Versus OnabotulinumtoxinA in the Treatment of Forehead Rhytides
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lupo Center for Aesthetic and General Dermatology (Other)
Collaborators: Evolus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pra vs Ona Spread 2023
Record Dates: First submitted 2023-03-09; First posted 2023-04-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Rhytides
Keywords: Rhytides; Prabotulinumtoxin A-xvfs; Onabotulinumtoxin A; Botox; Jeaveau; Neuromodulator; Frontalis
MeSH Terms: interventions — prabotulinumtoxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to have either their right forehead or left forehead treated with 4 units or 0.1 cc of prabotulinumtoxinA 2.5 cm above the orbital rim. As a control, the contralateral forehead half will receive 4 units or 0.1 cc of onabotulinumtoxinA at the same dilution at the same time.
Who Masked: Participant, Investigator
Masking Description: The left and right-side assignment will be determined based on the treating physician's selection of a sealed envelope using random numbers on the treatment day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental half (Experimental): Each subject will be randomized to have either their right forehead or left forehead treated with 4 units or 0.1 cc of prabotulinumtoxinA 2.5 cm above the orbital rim.
  Interventions: Drug: PrabotulinumtoxinA-Xvfs
- Comparator half (Active Comparator): Each subject will be randomized to have either their right forehead or left forehead treated with 4 units or 0.1 cc of onabotulinumtoxinA 2.5 cm above the orbital rim.
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: PrabotulinumtoxinA-Xvfs — All subjects will receive one injection of 4 units or 0.1 cc of prabotulinumtoxin A into the frontalis at a single point 2.5 cm above the orbital rim at the mid-pupillary line.
  The preparation of the 100-unit vial of prabotulinumtoxinA will be reconstituted gently and without shaking with 2.5 cc of 0.9% preserved normal saline solution. The investigator performing the injections will reconstitute study vials.
  Subjects will be injected intramuscularly using a hubless tuberculin syringe. Injections will be done at a 90-degree angle or perpendicular to the skin surface. The target sites will be the mid-line of the pupil and 2.5 cm above the orbital rim.
  Other Names: Jeaveau
  Arms: Experimental half
Drug: OnabotulinumtoxinA — All subjects will receive one injection of 4 units or 0.1 cc of onabotulinumtoxinA into the frontalis at a single point 2.5 cm above the orbital rim at the mid-pupillary line.
  The preparation of the 100-unit vial of onabotulinumtoxinA will be reconstituted gently and without shaking with 2.5 cc of 0.9% preserved normal saline solution. The investigator performing the injections will reconstitute study vials.
  Subjects will be injected intramuscularly using a hubless tuberculin syringe. Injections will be done at a 90-degree angle or perpendicular to the skin surface. The target sites will be the mid-line of the pupil and 2.5 cm above the orbital rim.
  Other Names: Botox
  Arms: Comparator half

SUMMARY:
Ten subjects will be enrolled in the study. Each subject will have their left and right forehead randomly assigned to receive 4 units of PrabotulinumtoxinA-xvfs or OnabotulinumtoxinA. Subjects will be reassessed at 2 weeks for evaluation of rhytide diminution around each injection point to assess relative diffusion of each drug in the forehead.

DETAILED DESCRIPTION:
This is a prospective, single-center, blinded, randomized, split-face study to investigate the area of spread or diffusion of onabotulinumtoxinA and prabotulinumtoxinA at the same dilution and dose in the treatment of forehead lines in adult subjects.

Ten adult subjects, 18 years or older, with moderate-to-severe dynamic and none-to-minimal static forehead lines will be enrolled. Upon enrollment and after a thorough review of the inclusion and exclusion criteria as well as obtaining written and informed consent, each subject will be randomized to have either their right forehead or left forehead treated with 4 units or 0.1 cc of prabotulinumtoxinA 2.5 cm above the orbital rim. As a control, the contralateral forehead half will receive 4 units or 0.1 cc of onabotulinumtoxinA at the same dilution. If applicable, a urine pregnancy test will be obtained prior to treatment. Subjects may be treated on the same day that they are screened and provide informed consent. Given the small volume of injection, tuberculin hubless syringes will be used to ensure accuracy of specific injection volumes. Injections will be delivered intramuscularly with the needle at a 90-degree angle or perpendicular to the skin surface. The left and right-side assignment will be determined based on the treating physician's selection of a sealed envelope using random numbers on the treatment day.

Following initial treatment, the subjects will be re-evaluated at a Day 14. Surface area of rhytide reduction will be measured in centimeters squared (incorporating length and width measurements) two-weeks post-injection to assess differences, if any, in rhytid reduction on each side of the forehead by a blinded investigator. The field of rhytid reduction (visual absence of horizontal forehead rhytids) will be measured while the frontalis fully contracted. Any adverse events will be recorded at the 2-week follow up. After the Day 14 assessment subjects will exit the study after which the investigator will assess the patient for any asymmetry and if the investigator deems it appropriate and the subject desires it, a touch up correction will be performed.

Subjects will be photographed at baseline and two weeks after treatment using Visia and 2D photography. Photos will be taken before and after marking the points of injection. Moreover, photos will be taken both with the frontalis muscle fully relaxed and fully contracted.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Moderate-to-severe dynamic forehead rhytides and none-to-minimal static forehead rhytides (score of 3 to 4 and score of 0 to 1, respectively, using a 5-point validated grading scale for forehead lines)1
* Subjects in good general health based on investigator's judgment and medical history
* Willingness to have facial exams and photos performed
* Must be willing to give and sign an informed consent form and photographic release form
* Negative urine pregnancy test result at the time of study entry (if applicable)
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Previous treatment with botulinum toxin of any serotype in the forehead area within the last 6 months
* History of permanent or long-acting fillers such as silicone, Sculptra® or Radiesse® in the treatment area
* Current history of substance abuse, including alcohol or other drugs
* Concurrent use of medications that affect neuromuscular transmission such as aminoglycoside antibiotics, anticholinesterases, lincosamides and polymyxins
* Marked facial asymmetry
* History of facial nerve palsy
* Medical condition that may affect neuromuscular function (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis)
* Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
* Known allergy or hypersensitivity to botulinum toxin preparation
* Any planned surgical intervention to the face for the duration of the trial
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* Subjects with tattoos or excessive scarring in the treatment areas
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Surface area of rhytid diminution | 14 days post-treatment
  Primary endpoint is surface area of rhytid diminution. Surface area of rhytid reduction will be measured in centimeters squared (incorporating length and width measurements) two-weeks post-injection to assess differences, if any, in rhytid reduction on each side of the forehead by the blinded investigator.

SECONDARY OUTCOMES:
5-point photonumeric scale for resting or static and hyperkinetic or dynamic horizontal forehead lines | 14 days post-treatment
  Change in 5-point photonumeric scale for resting or static and hyperkinetic or dynamic horizontal forehead lines: 0 = no wrinkles, 1 = minimal wrinkles, 2 = mild wrinkles, 3 = moderate wrinkles, 4 = severe wrinkles.
Adverse events | 14 days post-treatment
  Any adverse events will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Lupo Center for Aesthetic and General Dermatology, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carruthers A, Carruthers J, Hardas B, Kaur M, Goertelmeyer R, Jones D, Rzany B, Cohen J, Kerscher M, Flynn TC, Maas C, Sattler G, Gebauer A, Pooth R, McClure K, Simone-Korbel U, Buchner L. A validated grading scale for marionette lines. Dermatol Surg. 2008 Nov;34 Suppl 2:S167-72. doi: 10.1111/j.1524-4725.2008.34366.x. PMID 19021675
- [Background] Beer KR, Shamban AT, Avelar RL, Gross JE, Jonker A. Efficacy and Safety of PrabotulinumtoxinA for the Treatment of Glabellar Lines in Adult Subjects: Results From 2 Identical Phase III Studies. Dermatol Surg. 2019 Nov;45(11):1381-1393. doi: 10.1097/DSS.0000000000001903. PMID 30893162
- [Background] Lorenc ZP, Adelglass JM, Avelar RL, Baumann L, Beer KR, Cohen JL, Cox SE, Dayan SH, Dover JS, Downie JB, Draelos ZD, Goldman MP, Gross JE, Joseph JH, Kaufman-Janette J, Moy RL, Nestor M, Schlessinger J, Smith SR, Weiss RA. The Second of Two One-Year, Multicenter, Open-Label, Repeat-Dose, Phase II Safety Studies of PrabotulinumtoxinA for the Treatment of Moderate to Severe Glabellar Lines in Adult Patients. Aesthet Surg J. 2021 Nov 12;41(12):1423-1438. doi: 10.1093/asj/sjaa382. PMID 33944913
- [Background] Taylor SC, Grimes PE, Joseph JH, Jonker A, Avelar RL. PrabotulinumtoxinA for the Treatment of Moderate-to-Severe Glabellar Lines in Adult Patients With Skin of Color: Post Hoc Analyses of the US Phase III Clinical Study Data. Dermatol Surg. 2021 Apr 1;47(4):516-521. doi: 10.1097/DSS.0000000000002864. PMID 33165078
- [Background] Hsu TS, Dover JS, Arndt KA. Effect of volume and concentration on the diffusion of botulinum exotoxin A. Arch Dermatol. 2004 Nov;140(11):1351-4. doi: 10.1001/archderm.140.11.1351. PMID 15545544